CLINICAL TRIAL: NCT04564313
Title: Clinical Study of Anti-PD-1 Antibody Camrelizumab in the Treatment of Recurrent Hepatocellular Carcinoma After Liver Transplantation
Brief Title: Safety and Efficacy of Camrelizumab (Anti-PD-1 Antibody) in Recurrent HCC After Liver Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wang Guoying, M.D., Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2020]-02-061-01
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab treatment (Experimental): Camrelizumab (SHR-1210), 200mg, I.V., Q3W
  Interventions: Drug: Camrelizumab treatment

INTERVENTIONS:
Drug: Camrelizumab treatment — Camrelizumab (SHR-1210), 200mg, I.V., Q3W

SUMMARY:
This is a prospective clinical study to investigate the safety and efficacy of anti-PD-1 immunotherapy (Camrelizumab) in patients with recurrent hepatocellular carcinoma (HCC) after liver transplantation. All of the enrolled patients have a background of liver transplantation for HCC. Due to the tumor recurrence, patients are not suitable for curative surgical resection, and targeted therapy provides poor therapeutic effect, leading to tumor progression or intolerance. Before immunotherapy, the PD-L1 expression was confirmed negative in the graft liver by immunohistochemistry, and patients continued targeted therapy as part of a combined antitumor regimen. In addition, the immunosuppression schedule is also reduced to a low level.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, male or female;
2. Pathologically confirmed hepatocellular carcinoma after liver transplantation;
3. Tumor recurrence or metastasis is confirmed by CT and/or MRI examination, and neither intrahepatic recurrence nor extrahepatic metastasis is suitable for surgical resection;
4. At least one measurable recurrent or metastatic tumor lesion;
5. Tumor progression (mRECIST) or intolerance to treatment was assessed at least 1 month after oral administration of sorafenib or lenvatinib;
6. The expected survival time is more than 3 months;
7. Child-Pugh grade A or B (≤7 points);
8. Other vital organs' function: The absolute count of neutrophils ≥1.5×10E9/L; Platelet ≥50×10E9/L; Hemoglobin ≥9g/dL; Serum albumin ≥2.8g/dL; Thyroid stimulating hormone (TSH) ≤1 times ULN (If TSH is abnormal, T3 and T4 levels should be examined at the same time. Then, if both T3 and T4 levels are normal, patient could be enrolled); Bilirubin ≤1.5 times ULN; ALT and AST ≤3 times ULN; Serum creatinine ≤1.5 times ULN;
9. ECOG score 0-2 points;
10. Patients have sufficient understanding and voluntarily sign the informed consent, and are willing and able to comply with the visit, treatment plan, laboratory examination and other requirements of the study schedule.

Exclusion Criteria:

1. Positive PD-L1 expression in liver biopsy by immunohistochemistry (either liver parenchyma or non-parenchymal cells);
2. Be Allergic to Camrelizumab;
3. ≥ Grade II myocardial ischemia or myocardial infarction;
4. With hypertension that can't be controlled to normal level with medication (SBP >140mmHg, DBP >90mmHg);
5. With abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), and with a history of gastrointestinal bleeding within 6 months;
6. With high risk of bleeding or is receiving thrombolysis or anticoagulant therapy;
7. With autoimmune diseases including systemic lupus erythematosus, rheumatoid arthritis, psoriasis, etc;
8. The primary liver disease for liver transplantation was autoimmune hepatitis, primary biliary cirrhosis, or primary sclerosing cholangitis;
9. With pulmonary diseases such as interstitial pneumonia and poor lung function;
10. Participating in clinical trials of other experimental drugs within four weeks;
11. With infections requiring systemic treatment;
12. With positive infection of human immunodeficiency virus (HIV);
13. Special groups that not recommended in the instructions of Camrelizumab: with moderate or severe insufficiency of liver and renal function;
14. With MDM2/4 amplification, EGFR mutation, or JAK mutation by NGS sequencing;
15. With other factors that may influence the safety or compliance;
16. During the treatment of acute rejection or within 1 month after treatment;
17. Poor compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Objective Response Rate after Camrelizumab treatment according to the mRECIST

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Time from the initiation of Camrelizumab treatment to the patient death from any cause
Progression-free Survival (PFS) | 2 years
  Time from the initiation of Camrelizumab treatment to radiological tumor progression or death from any cause
Time to Progression (TTP) | 2 years
  Time from the initiation of Camrelizumab treatment to radiological tumor progression
Serious Adverse Event (SAE) | 2 years
  The incidence of serious adverse event caused by Camrelizumab treatment
Graft Rejection (GR) | 2 years
  The incidence of graft rejection during the Camrelizumab treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China